CLINICAL TRIAL: NCT04594265
Title: Weight-Adjusted Dosing of 3-OHB in Patients With Chronic Heart Failure
Acronym: KINETICS2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Kristian Hylleberg Christensen, MD, Aarhus University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KETO-KINETICS 2 1-10-72-23-20
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Heart Failure; Ketosis
Keywords: Hemodynamics
MeSH Terms: conditions — Heart Failure; Ketosis

STUDY DESIGN:
Intervention Model Description: Patients are studied in a randomized single-blind cross-over design.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ketone Monoester (Experimental): Weight-adjusted dose of 3-OHB Monoester (KetoneAID KE4, Virginia, US) 0.5 g/kg (max 50 g)
  Interventions: Dietary Supplement: KetoneAid KE4 Pro Monoester
- Placebo Treatment (Placebo Comparator): Maltodextrin-based placebo (Science In Sport, UK) in isocaloric dose to the experimental arm.
  Interventions: Dietary Supplement: Science in Sport Go Enegy
- Ketone Monoester in presence of low-dose insulin clamp (Active Comparator): Same as experimental arm, but in the presence of a low-dose insulin clamp to suppress free fatty acid metabolism
  Interventions: Dietary Supplement: KetoneAid KE4 Pro Monoester

INTERVENTIONS:
Dietary Supplement: KetoneAid KE4 Pro Monoester — A dietary supplement containing ketone monoester.
  Arms: Ketone Monoester; Ketone Monoester in presence of low-dose insulin clamp
Dietary Supplement: Science in Sport Go Enegy — Dosis isocaloric to the KetoneAid Arm
  Arms: Placebo Treatment

SUMMARY:
We aim to investigate the hemodynamic effects of weight-adjusted dosing of ketone monoester en patients with chronic heart failure.

ELIGIBILITY:
Inclusion criteria: Chronic HF: NYHA class II-III, left ventricular ejection fraction (LVEF) <40%

Exclusion Criteria: Diabetes or HbA1c >48 mmol/mol, significant cardiac valve disease, severe stable angina pectoris, severe comorbidity as judged by the investigator, inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Cardiac Output (L/min) | 3 hours - Area under the curve
  Change in Cardiac output measured by Swann-Ganz Catherization during study period,

SECONDARY OUTCOMES:
Left Ventricular Ejection Fraction | 3 hours - Area under the curve
  Change in LVEF measured by echocardiography during study periode
Blood Ketones | 3 hours
  Change in blood Ketones measured by venous blood samples
Blood pH | 3 hours
  Change in venous blood pH during the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No